CLINICAL TRIAL: NCT02761018
Title: Using Technology to Share Fitness Goals and Results to Improve Diabetes Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FWH20160062H
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fitness Tracker (Experimental): will use a fitness tracker but will not be able to see other participant's data
  Interventions: Behavioral: Fitness Tracker
- Fitness Tracker with Group Participation (Experimental): will use a fitness tracker and will be able to see other member's daily and weekly results
  Interventions: Behavioral: Behavioral: Fitness Tracker

INTERVENTIONS:
Behavioral: Behavioral: Fitness Tracker — will use a fitness tracker but will not be able to see other participant's data
  Arms: Fitness Tracker with Group Participation
Behavioral: Fitness Tracker — will use a fitness tracker and will be able to see other member's daily and weekly results
  Arms: Fitness Tracker

SUMMARY:
The investigators will recruit DoD beneficiaries, aged 18 years or older and diagnosed as being Type II diabetic. Patients will be randomized into one of two groups. Group 1 will use a fitness tracker but will not be able to see other participants data and group 2 will use a fitness tracker and will be able to see other members daily and weekly results. Outcome measures will be assessed at baseline, 3 months and 6 months to include hemoglobin A1c, weight, body mass index, blood pressure, and number of hours and days fitness tracker is used. The goal is to see if the group randomized into an online community will have improved activity and outcome measurements compared with those who use the pedometer alone.

DETAILED DESCRIPTION:
Male and female DoD beneficiaries ages 18 years or older who have been diagnosed with Type II diabetes, will be recruited at the Mike O'Callaghan Federal Medical Center (MOFMC).

Screening Visit:

* Obtain signed Informed Consent Document and HIPAA Authorization (research-driven).
* Record: Date of birth, phone number, age, gender, race, ethnicity, social security number, current email address, height (in inches), weight (in pounds), blood pressure, medications list including any over-the-counter and prescription weight loss medication (name, strength, dose) or supplements.
* Subjects will have the following standard of care blood test drawn which include:

  * Hemoglobin A1c via 1 venipuncture (5-10 mls, approximately 1-2 teaspoons of blood will be drawn)

Visit 1 (Day 1 within 1 week of Screening Visit):

* Record: Weight (in pounds), blood pressure, and any changes to their medications list.
* Subjects will complete the RAND 36 Item Health Survey.
* Subjects will complete the Intake Questionnaire.
* Subjects will be assigned their Fitness Tracker username and their username and password will be recorded by the Research Coordinator.
* Subjects will be given User Instructions based off of their randomization group.
* Subjects will be instructed to follow all research procedures and that failure to do so may result in the removal from the study and the return of the Fitness Tracker.
* Subjects will be randomized by the research coordinator using a random-number generator into one of two groups (research-driven):

  * Group 1: will use a fitness tracker but will not be able to see other participant's data.
  * Group 2: will use a fitness tracker and will be able to see other member's daily and weekly results.

    * Both groups will receive the scripted feedback at set time intervals by the Research Coordinators.
* Subjects will be provided a fitness tracker and instructed on how to use it.

  * If subject is a DoD beneficiary, and finishes all study-related procedures at month 6, they will keep the fitness tracker. If a subject does not complete all study-related procedures, they will be asked to return the fitness tracker so the investigators can erase their data and re-issue to another study subject.
  * If subject is active duty or a DoD employee, regardless of their study completion, they will be asked to complete Temporary Issue Receipt and bring back the fitness tracker at the end of the study.

Visit 2 (Month 3/90 days post Visit 1):

* Record: Weight (in pounds), blood pressure and any changes to their medications list.
* Subjects will complete the RAND 36 Item Health Survey.
* Subjects will complete the Follow up Questionnaire.
* Obtain information from their fitness tracker.
* Subjects will have the following standard of care blood test drawn which include:

  * Hemoglobin A1c via 1 venipuncture (5-10 mls, approximately 1-2 teaspoons of blood will be drawn)

Final Visit 3 (Month 6/90 days post Visit 2):

* Record: Weight (in pounds), blood pressure and any changes to their medications list.
* Subjects will complete the RAND 36 Item Health Survey and be asked some additional questions.
* Subjects will complete the Follow up Questionnaire.
* Obtain information from their fitness tracker.
* Subjects will have the following standard of care blood test drawn which include:

  * Hemoglobin A1c via 1 venipuncture (5-10 mls, approximately 1-2 teaspoons of blood will be drawn)

ELIGIBILITY:
YOU MUST BE ABLE TO GET CARE AT NELLIS AFB (A MILITARY INSTALLATION) IN ORDER TO PARTICIPATE IN THIS STUDY.

Inclusion:

* Male and female DoD beneficiaries, age 18 years or older, who have been diagnosed with Type II Diabetes
* Ability to set up fitness tracking software on personal computer or cell phone
* Ability to learn and use personal activity monitor

Exclusion:

* Male and female DoD beneficiaries, under the age of 18 years
* Unwilling to share personal fitness results anonymously
* Inability to do 4 metabolic equivalents of exercise (walk 100feet, walk up flight of stairs etc).
* Inability to walk without the use of assistive devices (cane is OK)
* Medical problem which would make walking unsafe (recent surgery, uncontrolled heart condition, fall risk etc).
* No special populations (e.g., pregnant women, children, prisoners, detainees) will be recruited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Reduction in hemoglobin a1c | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Carlsen, MD, Principal Investigator — Principal Investigator
Locations (1):
- Mike O'Callaghan Federal Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
we do not plan on sharing data